CLINICAL TRIAL: NCT04978493
Title: A Phase IIa, Randomised, Double-blind, Placebo-controlled Trial to Evaluate the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of BI 706321 Orally Administered for 12 Weeks in Patients With Crohn's Disease (CD) Receiving Ustekinumab Induction Treatment
Brief Title: A Study to Test Whether BI 706321 Combined With Ustekinumab Helps People With Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1425-0003; 2020-004527-16 (EudraCT Number)
Record Dates: First submitted 2021-07-26; First posted 2021-07-27 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Intervention Model Description: Ustekinumab treatment is open-label for the Sponsor, patients and investigator/site staff.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 706321 and ustekinumab (Experimental): Participants with moderately to severely active Crohn's Disease (CD) administered one dose of 8 milligram (mg) BI 706321 as tablets orally once per day in the morning for 12 weeks in conjunction with standard induction dosing of ustekinumab, followed by ustekinumab maintenance dosing for an additional 36 weeks.
  A single intravenous infusion of 260 mg ustekinumab (body weight ≤55 kilogram [kg]), 390 mg ustekinumab (body weight 55-85 kg), or 520 mg ustekinumab (body weight >85 kg) was administered on Day 0, followed by subcutaneous injection of 90 mg ustekinumab every 8 weeks.
  Interventions: Drug: BI 706321; Drug: Ustekinumab
- Placebo and ustekinumab (Placebo Comparator): Participants with moderately to severely active CD administered one dose of placebo matching BI 706321 as tablets orally once per day in the morning for 12 weeks in conjunction with standard induction dosing of ustekinumab, followed by ustekinumab maintenance dosing for an additional 36 weeks.
  A single intravenous infusion of 260 mg ustekinumab (body weight ≤55 kilogram [kg]), 390 mg ustekinumab (body weight 55-85 kg), or 520 mg ustekinumab (body weight >85 kg) was administered on Day 0, followed by subcutaneous injection of 90 mg ustekinumab every 8 weeks.
  Interventions: Drug: Ustekinumab; Drug: Placebo

INTERVENTIONS:
Drug: BI 706321 — One dose of 8 mg as tablets orally once per day in the morning
  Arms: BI 706321 and ustekinumab
Drug: Ustekinumab — A single intravenous infusion of 260 mg (body weight ≤55 kg), 390 mg (body weight 55-85 kg), or 520 mg (body weight >85 kg) was administered on Day 0, followed by subcutaneous injection of 90 mg every 8 weeks.
Drug: Placebo — One dose of placebo matching BI 706321 as tablets orally once per day in the morning
  Arms: Placebo and ustekinumab

SUMMARY:
This study is open to adults, aged 18-75 years, with moderate to severe Crohn's disease.

The purpose of this study is to find out whether BI 706321 combined with ustekinumab helps people with Crohn's disease. BI 706321 is a medicine being developed to treat Crohn's disease. Ustekinumab is a medicine already used to treat Crohn's disease.

Participants are put into 2 groups randomly, which means by chance. One group gets BI 706321 and ustekinumab. The other group gets placebo and ustekinumab.

Participants take BI 706321 or placebo as tablets every day. Placebo tablets look like BI 706321 tablets but do not contain any medicine. Ustekinumab is given as an infusion into a vein once at the beginning of the study. After that, ustekinumab is given as an injection under the skin every 2 months. Participants take BI 706321 or placebo in combination with ustekinumab for 3 months. After that, participants receive only ustekinumab for another 9 months.

Participants are in the study for about 1 year. During this time, they visit the study site about 13 times. At 3 of the visits, doctors do a colonoscopy to examine the bowel. The results from the colonoscopies are compared between the 2 groups. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn Disease (CD) for at least 3 months prior to visit 1, as confirmed at any time in the past by endoscopy and/OR, radiology, and supported by histology.
* Elevated C-reactive protein (≥ 5 mg/L) OR elevated fecal calprotectin (≥ 250 µg/g)
* Symptomatic CD defined as Crohn's Disease Activity Index (CDAI) ≥150.
* Presence of mucosal ulcers in at least one segment of the ileum or colon and a Simple Endoscopic Score for Crohn's disease (SES-CD) score ≥ 7 (for patients with isolated ileitis ≥4).
* Patients who are experienced at least 1 tumor necrosis factor (TNF) antagonists at a dose approved for CD. Patients may have stopped TNF antagonist treatment due to primary or secondary non-responsiveness, intolerance, or for other reasons.
* May be receiving a therapeutic dose of the following:

  * Oral 5-aminosalicylic acid (5-ASA) compounds must have been at a stable dose for at least 4 weeks prior to randomisation and must continue on this dose until week 12 and/or
  * Oral corticosteroids if indicated for treatment of CD must be at a prednisone equivalent dose of ≤ 20 mg/day, or ≤ 9 mg/day of budesonide, and have been at a stable dose for at least 2 weeks immediately prior to randomisation and must continue on this dose until week 12. and/or
  * Azathioprine (AZA), mercaptopurine (MP), or methotrexate (MTX), provided that dose has been stable for the 8 weeks immediately prior to randomisation and must continue on this dose until week 12.
* Women of childbearing potential must be ready and able to use highly effective methods of birth control.
* Further inclusion criteria apply

Exclusion Criteria:

* Have any current or prior abscesses, unless they have been drained and treated at least 6 weeks prior to randomisation and are not anticipated to require surgery. Patients with active fistulas may be included if there is no anticipation of a need for surgery and there are currently no abscesses present based on investigator's judgement.
* Have complications of CD such as strictures, stenosis, short bowel syndrome, or any other manifestation that might require surgery, or could preclude the use of SES-CD/CDAI to assess response to therapy, or would possibly confound the evaluation of benefit from treatment with BI 706321 (based on investigator's judgement).
* Patient with an inflammatory bowel disease (IBD) diagnosis other than CD.
* Have had any kind of bowel resection or diversion within 4 months or any other intra-abdominal surgery within 3 months prior to visit 1. Patients with current ileostomy, colostomy, or ileorectal anastomosis are excluded.
* Treatment with:

  * Any non-biologic medication for IBD (e.g.tacrolimus or mycophenolate mofetil, systemic corticosteroids), other than those allowed per inclusion criteria, within 30 days prior to randomisation
  * Any biologic treatment with a TNF-alpha antagonist (adalimumab, infliximab, golimumab, certolizumab pegol) or vedolizumab (or a biosimilar of these drugs) within 4 weeks prior to randomisation. (If drug level testing for previously used biologic treatment confirms no detectable drug level before randomisation, patient can be enrolled despite not having completed 4 week from last treatment.)
  * Any previous treatment with ustekinumab (or a biosimilar of this drug)
  * Any previous treatment with an investigational (or subsequently approved) non-biologic/biologic drug for CD (including but not limited to JAK inhibitors [e.g. upadacitinib], S1P modulators, IL-23 inhibitors [e.g. risankizumab], antiintegrins).
  * Any investigational drug for an indication other than CD during the course of the actual study and within 30 days or 5 half-lives (whichever is longer) prior to randomisation.
  * Any prior exposure to rituximab within 1 year prior to randomisation.
* Positive stool examination for C difficile or other intestinal pathogens <30 days prior to randomization
* Evidence of colonic moderate/severe mucosal dysplasia or colonic adenomas, unless properly removed
* Increased risk of infectious complications (e.g. recent pyogenic infection, any congenital or acquired immunodeficiency (e.g. human immunodeficiency virus (HIV)), past organ or stem cell transplantation (with exception of a corneal transplant > 12 weeks prior to screening) or have ever received stem cell therapy (e.g., Prochymal). Prior treatment with a somatic cell therapy product (e.g., Alofisel) is not excluded, provided it was administered > 8 weeks prior to randomisation.
* Live or attenuated vaccination within 4 weeks prior to randomisation.
* Presence of clinically significant acute or chronic infections not otherwise listed, including viral hepatitis, COVID-19, or others based on investigator's judgement.
* A marked baseline prolongation of QT/QTc interval (such as QTcF intervals that are greater than 450 ms for men, 470 ms for female) or any other relevant electrocardiogram (ECG) finding at screening. Both have to be confirmed by repeated ECG recording.
* Further exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-08-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (15):
  - California Medical Research Associates Inc., Northridge, California
  - Sweet Hope Research Specialty Inc, Hialeah, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - I.H.S Health, LLC, Kissimmee, Florida
  - Advanced Research Institute, Inc., Orlando, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - BVL Clinical Research, Liberty, Missouri
  - Carolina Digestive Diseases, Greenville, North Carolina
  - Houston Methodist Hospital, Houston, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - GI Alliance, Southlake, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
- Belgium (6):
  - Brussels - UNIV St-Pierre, Brussels
  - AZ Maria Middelares, Ghent
  - AZ Sint-Lucas - Campus Sint Lucas, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
  - UNIV Ambroise Paré, Mons
- Czechia (2):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - University Hospital Ostrava, Ostrava
- Aalborg Sygehus Syd, Aalborg, Denmark
- Universitätsklinikum Ulm, Ulm, Germany
- Hungary (3):
  - Clinexpert Kft., Budapest
  - University of Debrecen Clinical Centre, Debrecen
  - Bugat Pal Hospital, Gyongyos, Gyöngyös
- Italy (7):
  - Policlinico Universitario Mater Domini, Universita di Catanzaro, Catanzaro
  - IRCCS Fondazione Ospedale Maggiore, Milan
  - IRCCS San Raffaele, Milan
  - Osp.Sacro Cuore-Don Calabria, Negrar (VR)
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Az. Ospedaliera Universitaria Polic.Tor Vergata, Roma
  - IRCCS Policlinico San Donato, San Donato Milanese (MI)
- Netherlands (2):
  - Radboud Universitair Medisch Centrum, Nijmegen
  - St Elisabeth Ziekenhuis, Tilburg
- Poland (6):
  - NZOZ Medical Center KERmed, Bydgoszcz
  - Indywidualna Specjalistyczna Praktyka Lekarska Maciej Zymla, Knurów
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska sp. j., Ksawerów
  - Healthcare Center Gastromed - SCANMED GROUP, Lublin
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - National Medical Institute MSWiA, Warsaw
- Spain (5):
  - payee-Hospital Universitario Reina Sofia. Cordoba, Córdoba
  - Hospital La Princesa, Madrid
  - CEIC Corporacio Sanitaria Parc Taulí, Sabadell
  - Hospital Virgen Macarena, Seville
  - Hospital Politècnic La Fe, Valencia
- Royal Liverpool University Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase IIa, randomised, double-blind, placebo-controlled evaluation of male and female patients with Crohn's Disease (CD), using BI 706321 therapy in combination with a backbone ustekinumab induction regimen.
Pre-assignment Details: Subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) met all inclusion and no exclusion criteria. Subjects were not to be allocated to a treatment group if any entry criteria were violated. Subjects signed and dated an informed consent form according to local regulatory and legal requirements, and were informed that they were free to withdraw their consent at any time without penalty or prejudice.
Period: Overall Study
Arm/Group | BI 706321 and Ustekinumab | Placebo and Ustekinumab
Started | 24 | 25
Completed (Number of participants who completed the 12-weeks treatment with BI 706321 or placebo) | 23 | 24
Not Completed | 1 | 1
Not completed — No reason available | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): all randomized patients who received at least 1 dose of trial medication and have analyzable post-baseline data (observed or imputed) in at least 1 efficacy/biological/histological parameter.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 706321 and Ustekinumab | Placebo and Ustekinumab | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.8 (14.9) | 47.8 (13.8) | 43.4 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 21 | 25 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 22 | 22 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Simple Endoscopic Score for Crohn's disease (SES-CD) [Mean (Standard Deviation); unit: Score on a scale] — The SES-CD is a numerical grading system composed of 4 variables (presence of ulcers, ulcerated surface, affected surface, presence of narrowings) recorded sequentially in 5 segments: rectum, left colon, transverse colon, right colon, ileum. Each variable is assigned a value from 0 to 3, and the total score, ranging from 0 to 56, is obtained by adding each variable. Higher values indicate worse endoscopic inflammation. To achieve a score of 56, the maximum score for the "presence of narrowings" variable has to be be 2 (not 3) for the four segments leading up to the ileum.
  Score on a scale | 14.1 (5.8) | 12.0 (4.9) | 13.0 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Simple Endoscopic Score for Crohn's Disease (SES-CD) at Week 12
Description: Absolute change from baseline in Simple Endoscopic Score for Crohn's disease (SES-CD) at Week 12 is reported. The SES-CD is a numerical grading system composed of 4 variables (presence of ulcers, ulcerated surface, affected surface, presence of narrowings) recorded sequentially in 5 segments: rectum, left colon, transverse colon, right colon, ileum. Each variable is assigned a value from 0 to 3, and the total score, ranging from 0 to 56, is obtained by adding each variable. Higher values indicate worse endoscopic inflammation. To achieve a score of 56, the maximum score for the "presence of narrowings" variable has to be be 2 (not 3) for the four segments leading up to the ileum. The analysis was a restricted maximum likelihood (REML) based analysis of covariance (ANCOVA). For the ANCOVA model, absolute change in SES-CD score was the dependent variable, treatment group and baseline corticosteroid use (yes/no) were fixed effects and baseline SES-CD score was a continuous covariate.
Time Frame: Within 28 days before randomization (baseline) and 12 weeks after first drug administration.
Population: Full analysis set (FAS): all randomized patients who received at least 1 dose of trial medication and have analyzable post-baseline data (observed or imputed) in at least 1 efficacy/biological/histological parameter. If a subject discontinued after 6 weeks and had an assessment during the Week 8 visit window, the change in SES-CD score at Week 8 was carried forward to the Week 12 time point and used. If there was no post-baseline endoscopic assessment, baseline value was carried forward.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | BI 706321 and Ustekinumab | Placebo and Ustekinumab
Number analyzed (Participants) | 24 | 25
Score on a scale | -1.69 [-3.75 to 0.37] | -3.62 [-5.63 to -1.60]
Statistical Analysis 1: Comparison: BI 706321 and Ustekinumab vs Placebo and Ustekinumab; The analysis was a restricted maximum likelihood (REML) based analysis of covariance (ANCOVA). For the ANCOVA model, absolute change in SES-CD score was the dependent variable, treatment group and baseline corticosteroid use (yes/no) were fixed effects and baseline SES-CD score was a continuous covariate; Test type: Other; Difference of adjusted means = 1.92, 95% CI 2-sided [-0.99 to 4.84], Standard Error of Mean 1.45 — (Adjusted mean BI 706321 and ustekinumab) - (adjusted mean Placebo and ustekinumab)

2. Secondary Outcome: Percent Change in SES-CD From Baseline at Week 12
Description: Percent change in Simple Endoscopic Score for Crohn's disease (SES-CD) from baseline at Week 12 is reported. The SES-CD is a numerical grading system composed of 4 variables (presence of ulcers, ulcerated surface, affected surface, presence of narrowings) recorded sequentially in 5 segments: rectum, left colon, transverse colon, right colon, ileum. Each variable is assigned a value from 0 to 3, and the total score, ranging from 0 to 56, is obtained by adding each variable. Higher values indicate worse endoscopic inflammation. To achieve a score of 56, the maximum score for the "presence of narrowings" variable has to be be 2 (not 3) for the four segments leading up to the ileum. The analysis was a restricted maximum likelihood (REML) based analysis of covariance (ANCOVA). For the ANCOVA model, absolute change in SES-CD score was the dependent variable, treatment group and baseline corticosteroid use (yes/no) were fixed effects and baseline SES-CD score was a continuous covariate.
Time Frame: Within 28 days before randomization (baseline) and 12 weeks after first drug administration.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | BI 706321 and Ustekinumab | Placebo and Ustekinumab
Number analyzed (Participants) | 24 | 25
Percent change | -14.18 [-30.30 to 1.95] | -27.52 [-43.30 to -11.73]
Statistical Analysis 1: Comparison: BI 706321 and Ustekinumab vs Placebo and Ustekinumab; [analysis description as in outcome 1, analysis 1]; Test type: Other; Difference of adjusted means = 13.34, 95% CI 2-sided [-9.46 to 36.14], Standard Error of Mean 11.32 — (Adjusted mean BI 706321 and ustekinumab) - (adjusted mean Placebo and ustekinumab)

3. Secondary Outcome: Percentage of Patients With Endoscopic Response (Defined as >50% SES-CD Reduction From Baseline, or for an Induction Baseline SES-CD of 4, at Least a 2 Point Reduction From Induction Baseline) at Week 12
Description: Percentage of patients with endoscopic response (defined as >50% Simple Endoscopic Score for Crohn's disease (SES-CD) reduction from baseline, or for an induction baseline SES-CD of 4, at least a 2 point reduction from induction baseline) at Week 12 is reported. The SES-CD is a numerical grading system composed of 4 variables (presence of ulcers, ulcerated surface, affected surface, presence of narrowings) recorded sequentially in 5 segments: rectum, left colon, transverse colon, right colon, ileum. Each variable is assigned a value from 0 to 3, and the total score, ranging from 0 to 56, is obtained by adding each variable. Higher values indicate worse endoscopic inflammation. To achieve a score of 56, the maximum score for the "presence of narrowings" variable has to be be 2 (not 3) for the four segments leading up to the ileum. The method to provide confidence intervals for single proportions is based on the Wilson method.
Time Frame: Within 28 days before randomization (baseline) and 12 weeks after first drug administration.
Population: Full analysis set (FAS): all randomized patients who received at least 1 dose of trial medication and have analyzable post-baseline data (observed or imputed) in at least 1 efficacy/biological/histological parameter. If there were data at visits before and after one with a missing outcome, data was imputed as success only if both neighboring visits represented a success, independently of whether the before and after observations were selected for analysis based on the pre-defined time windows.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | BI 706321 and Ustekinumab | Placebo and Ustekinumab
Number analyzed (Participants) | 24 | 25
Percentage of patients | 12.5 [4.3 to 31.0] | 40.0 [23.4 to 59.3]
Statistical Analysis 1: Comparison: BI 706321 and Ustekinumab vs Placebo and Ustekinumab; Unadjusted risk difference between treatment groups were calculated simply as the difference in the observed percentage of patients. The method to provide confidence intervals for the unadjusted risk differences was derived from the Newcombe method; Test type: Other; Unadjusted risk difference = -27.50, 95% CI 2-sided [-48.42 to -2.64] — BI 706321 and ustekinumab - Placebo and ustekinumab

4. Secondary Outcome: Percentage of Patients With Endoscopic Response (Defined as >50% SES-CD Reduction From Baseline, or for an Induction Baseline SES-CD of 4, at Least a 2 Point Reduction From Induction Baseline) at Week 48
Description: Percentage of patients with endoscopic response (defined as >50% Simple Endoscopic Score for Crohn's disease (SES-CD) reduction from baseline, or for an induction baseline SES-CD of 4, at least a 2 point reduction from induction baseline) at Week 48 is reported. The SES-CD is a numerical grading system composed of 4 variables (presence of ulcers, ulcerated surface, affected surface, presence of narrowings) recorded sequentially in 5 segments: rectum, left colon, transverse colon, right colon, ileum. Each variable is assigned a value from 0 to 3, and the total score, ranging from 0 to 56, is obtained by adding each variable. Higher values indicate worse endoscopic inflammation. To achieve a score of 56, the maximum score for the "presence of narrowings" variable has to be be 2 (not 3) for the four segments leading up to the ileum. The method to provide confidence intervals for single proportions is based on the Wilson method.
Time Frame: Within 28 days before randomization (baseline) and 48 weeks after first drug administration.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | BI 706321 and Ustekinumab | Placebo and Ustekinumab
Number analyzed (Participants) | 24 | 25
Percentage of patients | 16.7 [6.7 to 35.9] | 16.0 [6.4 to 34.7]
Statistical Analysis 1: Comparison: BI 706321 and Ustekinumab vs Placebo and Ustekinumab; [analysis description as in outcome 3, analysis 1]; Test type: Other; Unadjusted risk difference = 0.67, 95% CI 2-sided [-20.49 to 22.12] — BI 706321 and ustekinumab - Placebo and ustekinumab

5. Secondary Outcome: Percentage of Patients With Endoscopic Remission (Defined as SES-CD Score of ≤2) at Week 12
Description: Percentage of patients with endoscopic remission (defined as Simple Endoscopic Score for Crohn's disease (SES-CD) score of ≤2) at Week 12 is reported. The SES-CD is a numerical grading system composed of 4 variables (presence of ulcers, ulcerated surface, affected surface, presence of narrowings) recorded sequentially in 5 segments: rectum, left colon, transverse colon, right colon, ileum. Each variable is assigned a value from 0 to 3, and the total score, ranging from 0 to 56, is obtained by adding each variable. Higher values indicate worse endoscopic inflammation. To achieve a score of 56, the maximum score for the "presence of narrowings" variable has to be be 2 (not 3) for the four segments leading up to the ileum. The method to provide confidence intervals for single proportions is based on the Wilson method.
Time Frame: 12 weeks after first drug administration.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | BI 706321 and Ustekinumab | Placebo and Ustekinumab
Number analyzed (Participants) | 24 | 25
Percentage of patients | 4.2 [0.7 to 20.2] | 8.0 [2.2 to 25.0]
Statistical Analysis 1: Comparison: BI 706321 and Ustekinumab vs Placebo and Ustekinumab; [analysis description as in outcome 3, analysis 1]; Test type: Other; Unadjusted risk difference = -3.83, 95% CI 2-sided [-21.14 to 13.25] — BI 706321 and ustekinumab - Placebo and ustekinumab

6. Secondary Outcome: Percentage of Patients With Endoscopic Remission (Defined as SES-CD Score of ≤2) at Week 48
Description: Percentage of patients with endoscopic remission (defined as Simple Endoscopic Score for Crohn's disease (SES-CD) score of ≤2) at Week 48 is reported. The SES-CD is a numerical grading system composed of 4 variables (presence of ulcers, ulcerated surface, affected surface, presence of narrowings) recorded sequentially in 5 segments: rectum, left colon, transverse colon, right colon, ileum. Each variable is assigned a value from 0 to 3, and the total score, ranging from 0 to 56, is obtained by adding each variable. Higher values indicate worse endoscopic inflammation. To achieve a score of 56, the maximum score for the "presence of narrowings" variable has to be be 2 (not 3) for the four segments leading up to the ileum. The method to provide confidence intervals for single proportions is based on the Wilson method.
Time Frame: 48 weeks after first drug administration.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | BI 706321 and Ustekinumab | Placebo and Ustekinumab
Number analyzed (Participants) | 24 | 25
Percentage of patients | 8.3 [2.3 to 25.8] | 8.0 [2.2 to 25.0]
Statistical Analysis 1: Comparison: BI 706321 and Ustekinumab vs Placebo and Ustekinumab; [analysis description as in outcome 3, analysis 1]; Test type: Other; Unadjusted risk difference = 0.33, 95% CI 2-sided [-17.67 to 18.78] — BI 706321 and ustekinumab - Placebo and ustekinumab

7. Secondary Outcome: Percentage of Patients With Biological Remission, Defined as C-Reactive Protein (CRP) < 5 mg/L and Faecal Calprotectin (FCP) < 250 ug/g at Week 12
Description: Percentage of patients with biological remission, defined as C-Reactive Protein (CRP) < 5 mg/L and faecal calprotectin (FCP) < 250 ug/g at Week 12 is reported. The method to provide confidence intervals for single proportions is based on the Wilson method.
Time Frame: 12 weeks after first drug administration.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | BI 706321 and Ustekinumab | Placebo and Ustekinumab
Number analyzed (Participants) | 24 | 25
Percentage of patients | 16.7 [6.7 to 35.9] | 20.0 [8.9 to 39.1]
Statistical Analysis 1: Comparison: BI 706321 and Ustekinumab vs Placebo and Ustekinumab; [analysis description as in outcome 3, analysis 1]; Test type: Other; Unadjusted risk difference = -3.33, 95% CI 2-sided [-24.91 to 18.85] — BI 706321 and ustekinumab - Placebo and ustekinumab

8. Secondary Outcome: Percentage of Patients With Biological Remission, Defined as C-Reactive Protein (CRP) < 5 mg/L and Faecal Calprotectin (FCP) < 250 ug/g at Week 48
Description: Percentage of patients with biological remission, defined as C-Reactive Protein (CRP) < 5 mg/L and faecal calprotectin (FCP) < 250 ug/g at Week 48 is reported. The method to provide confidence intervals for single proportions is based on the Wilson method.
Time Frame: 48 weeks after first drug administration.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | BI 706321 and Ustekinumab | Placebo and Ustekinumab
Number analyzed (Participants) | 24 | 25
Percentage of patients | 12.5 [4.3 to 31.0] | 16.0 [6.4 to 34.7]
Statistical Analysis 1: Comparison: BI 706321 and Ustekinumab vs Placebo and Ustekinumab; [analysis description as in outcome 3, analysis 1]; Test type: Other; Unadjusted risk difference = -3.50, 95% CI 2-sided [-23.86 to 17.34] — BI 706321 and ustekinumab - Placebo and ustekinumab

9. Secondary Outcome: Percentage of Patients With Clinical Remission at Week 12, Defined as a Crohn's Disease Activity Index (CDAI) Score of <150
Description: Percentage of patients with clinical remission at Week 12, defined as a Crohn's Disease Activity Index (CDAI) score of <150 is reported. The CDAI is comprised of eight variables which are summed after adjustment with a weighting factor, and the total score ranges from 0 to approximately 600, with higher scores indicating more severe disease. For certain variables (daily number of liquid or very soft stools, daily abdominal pain, daily general well-being, fever over 37.8 Celsius, taking medication for diarrhea) the average over 7 days was taken. The method to provide confidence intervals for single proportions is based on the Wilson method.
Time Frame: Data was collected for 7 days prior to 12 weeks after first drug administration.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | BI 706321 and Ustekinumab | Placebo and Ustekinumab
Number analyzed (Participants) | 24 | 25
Percentage of patients | 37.5 [21.2 to 57.3] | 56.0 [37.1 to 73.3]
Statistical Analysis 1: Comparison: BI 706321 and Ustekinumab vs Placebo and Ustekinumab; [analysis description as in outcome 3, analysis 1]; Test type: Other; Unadjusted risk difference = -18.50, 95% CI 2-sided [-42.32 to 8.89] — BI 706321 and ustekinumab - Placebo and ustekinumab

10. Secondary Outcome: Percentage of Patients With Clinical Remission at Week 48, Defined as a CDAI Score of <150
Description: Percentage of patients with clinical remission at Week 48, defined as a CDAI score of <150 is reported. The CDAI is comprised of eight variables which are summed after adjustment with a weighting factor, and the total score ranges from 0 to approximately 600, with higher scores indicating more severe disease. For certain variables (daily number of liquid or very soft stools, daily abdominal pain, daily general well-being, fever over 37.8 Celsius, taking medication for diarrhea) the average over 7 days was taken. The method to provide confidence intervals for single proportions is based on the Wilson method.
Time Frame: Data was collected for 7 days prior to 48 weeks after first drug administration.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | BI 706321 and Ustekinumab | Placebo and Ustekinumab
Number analyzed (Participants) | 24 | 25
Percentage of patients | 20.8 [9.2 to 40.5] | 20.0 [8.9 to 39.1]
Statistical Analysis 1: Comparison: BI 706321 and Ustekinumab vs Placebo and Ustekinumab; [analysis description as in outcome 3, analysis 1]; Test type: Other; Unadjusted risk difference = 0.83, 95% CI 2-sided [-21.53 to 23.41] — BI 706321 and ustekinumab - Placebo and ustekinumab

11. Secondary Outcome: Percentage of Patients With Clinical Response at Week 12, Defined by a CDAI Reduction From Baseline of at Least 100 Points, or a CDAI Score of <150
Description: Percentage of patients with clinical response at Week 12, defined by a CDAI reduction from baseline of at least 100 points, or a CDAI score of <150 is reported. The CDAI is comprised of eight variables which are summed after adjustment with a weighting factor, and the total score ranges from 0 to approximately 600, with higher scores indicating more severe disease. For certain variables (daily number of liquid or very soft stools, daily abdominal pain, daily general well-being, fever over 37.8 Celsius, taking medication for diarrhea) the average over 7 days was taken. The method to provide confidence intervals for single proportions is based on the Wilson method.
Time Frame: Within 28 days before randomization (baseline) and for 7 days prior to 12 weeks after first drug administration.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | BI 706321 and Ustekinumab | Placebo and Ustekinumab
Number analyzed (Participants) | 24 | 25
Percentage of patients | 45.8 [27.9 to 64.9] | 68.0 [48.4 to 82.8]
Statistical Analysis 1: Comparison: BI 706321 and Ustekinumab vs Placebo and Ustekinumab; [analysis description as in outcome 3, analysis 1]; Test type: Other; Unadjusted risk difference = -22.17, 95% CI 2-sided [-45.42 to 5.19] — BI 706321 and ustekinumab - Placebo and ustekinumab

12. Secondary Outcome: Number of Patients With Treatment-emergent Adverse Event (TEAE) Through End of Treatment (EoT) and the REP Period
Description: Number of patients with treatment-emergent adverse event (TEAE) through end of treatment (EoT) and the REP period is reported.
Time Frame: From first drug administration until 16 days after last drug administration, up to 27 weeks.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BI 706321 and Ustekinumab | Placebo and Ustekinumab
Number analyzed (Participants) | 24 | 25
Participants | 11 | 12

ADVERSE EVENTS:
Time Frame: From first drug administration, until end of follow-up period, up to 48 weeks.
Description: Full analysis set (FAS): all randomized patients who received at least 1 dose of trial medication and have analyzable post-baseline data (observed or imputed) in at least 1 efficacy/biological/histological parameter.
Arm/Group | BI 706321 and Ustekinumab | Placebo and Ustekinumab
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/24 | 1/25
Other Adverse Events (participants affected / at risk) | 0/24 | 6/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 706321 and Ustekinumab (N=24) | Placebo and Ustekinumab (N=25)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 706321 and Ustekinumab (N=24) | Placebo and Ustekinumab (N=25)
Vertigo (Ear and labyrinth disorders) | 0 | 2
Fatigue (General disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2
Rhinitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Due to trial discontinuation, patients that were ongoing in the follow-up period could not receive ustekinumab for the full 36 weeks, so End of Study assessments were either performed earlier or were missing, as was the case for endoscopies. Consequently, more patients had missing 48-week data that necessitated imputation via Non-response imputation or Last observation carried forward than there would have been had the trial continued as planned, so 48-week data must be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT04978493/Prot_002.pdf
  • Statistical Analysis Plan (2024-08-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT04978493/SAP_001.pdf